CLINICAL TRIAL: NCT07074925
Title: Video-Assisted Informed Consent for Neonatal Lumbar Puncture
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Texas at Austin (Other)
Responsible Party: Principal Investigator, Lina Palomares, Project Manager, University of Texas at Austin
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 00004883
Record Dates: First submitted 2025-07-01; First posted 2025-07-20 (Actual); Last update posted 2025-07-20 (Actual); Status verified 2025-07

CONDITIONS: Lumbar Puncture; Pediatrics; Emergency Department Patient; Informed Consent

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Video assisted consent (Experimental): The intervention group (n=50) will receive procedure information via a video explanation. The 2-minute video (available in English or Spanish) will use animation to explain the neonatal LP procedure, benefits, and risks.
  Interventions: Other: Video assisted informed consent
- Standard consent (Active Comparator): The control group (n=50) will receive standard procedure explanation.
  Interventions: Other: Standard consent

INTERVENTIONS:
Other: Video assisted informed consent — The 2-minute video (available in English or Spanish) will use animation to explain the neonatal LP procedure, benefits, and risks.
  Arms: Video assisted consent
Other: Standard consent — The standard consent group will receive usual procedure description and consent.
  Arms: Standard consent

SUMMARY:
The purpose of this study is to explore the effectiveness of video-assisted neonatal lumbar puncture consent processes against a conventional consent discussion to inform parents about pediatric lumbar puncture in the pediatric ED. We hypothesize that having a visual aid in addition to the verbal information presented in the consent process will lead to increased parent comprehension, decision-making, and satisfaction with the consent process. Furthermore, the findings from this study may have broader implications for improving the informed consent process for other medical procedures and interventions in pediatric settings.

DETAILED DESCRIPTION:
A neonatal lumbar puncture (LP), also known as a spinal tap, is a critical diagnostic procedure for detecting and managing serious infections such as meningitis in newborns. Ensuring that parents and caregivers fully understand the procedure, its risks, and its benefits is an essential aspect of the informed consent process. Traditionally, healthcare providers have relied on verbal and written methods to communicate this information to parents, aiming to facilitate comprehension and obtain consent for the procedure. However, there is growing evidence that these traditional methods may not always be sufficient in providing parents with a comprehensive understanding of the procedure, which could potentially impact the decision-making process and overall satisfaction with the care provided. After conventional consent discussions, parents are still often not aware of what the procedure will entail, the risks, how long the procedure will take, and what outcomes to expect. Language barriers can also contribute to misunderstandings during the consent process, even with the assistance of translation services.

Despite the importance of obtaining informed consent for neonatal LPs, there is a notable lack of research on the effectiveness of alternative methods for communicating this information, such as video-assisted consent. Video-based interventions have been shown to improve patient understanding and satisfaction in other medical contexts and may provide a more engaging and easily accessible means of conveying complex information related to the neonatal lumbar puncture procedure. Integrating video-assisted consent into the process could potentially enhance parent comprehension, decision-making, and satisfaction with the consent process.

The purpose of this study is to explore the effectiveness of video-assisted neonatal lumbar puncture consent processes against a conventional consent discussion to inform parents about pediatric lumbar puncture in the pediatric ED. We hypothesize that having a visual aid in addition to the verbal information presented in the consent process will lead to increased parent comprehension, decision-making, and satisfaction with the consent process. Furthermore, the findings from this study may have broader implications for improving the informed consent process for other medical procedures and interventions in pediatric settings.

A video-assisted informed consent intervention will be implemented in the Dell Children's Medical Center (DCMC) Emergency Department (ED). Parents whose children are recommended for LP will be randomly selected to receive either standard informed consent procedures or video-assisted informed consent. We plan to enroll 100 participants. The intervention group (n=50) will receive procedure information via a video and the control group (n=50) will receive standard procedure explanation. The 2-minute video (available in English or Spanish) will use animation to explain the neonatal LP procedure, benefits, and risks.

All participants will complete brief knowledge surveys after the intervention and will be asked to provide feedback on their satisfaction with the informed consent process. Pediatric emergency medicine physicians at Dell Children's collaborated to create the knowledge surveys using the Delphi method. The primary outcome to be assessed is the efficacy of the video intervention on parents' comprehension compared to the conventional discussion. Secondary outcomes will focus on parental satisfaction with the informed consent process and the rate of consent refusal.

ELIGIBILITY:
Inclusion Criteria:

* Children, age 0-7 months old who are recommended for lumbar puncture procedure during an ED visit.
* Caregiver fluent in English or Spanish

Exclusion Criteria:

* Previous enrollment in the study, i.e., the patient has been previously part of the current LP study. This will be confirmed by the study coordinator, PI, or co-I.
* Parent/guardian unwilling to complete surveys

Ages: 0 Months to 7 Months | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 100 (Estimated)
Dates: Start 2023-10-01 (Actual); Primary Completion 2024-11-15 (Actual); Study Completion 2025-11-15 (Estimated)

PRIMARY OUTCOMES:
Comprehension efficacy | Day 1
  Efficacy of the video intervention on parents' comprehension compared to the conventional consent discussion of the lumbar puncture procedure. Using the Delphi method, a knowledge survey was designed. The survey consists of 10 questions about the lumbar puncture procedure that are discussed in both the standard consent discussion and in the video. Each question has one correct response. The investigators will compare correct responses (individual questions and aggregate scores) between the two groups. The survey will be given to the parents/caregivers immediately after the procedure informed consent process.

SECONDARY OUTCOMES:
Parental satisfaction | Day 1
  Parental satisfaction of the consent process will be obtained using a single question with a Likert scale response option: "How satisfied were you with the consent process for the lumbar puncture procedure? Were you: very satisfied, satisfied, neither satisfied nor dissatisfied, dissatisfied, very dissatisfied." This question is part of a survey that will be given to parents/caregivers immediately after the consent process for the lumbar puncture procedure. Parents/caregivers of both groups will be asked this question and satisfaction ratings of the groups will be compared.

CONTACTS AND LOCATIONS:
Overall Officials: Matthew Wilkinson, MD, MPH, Study Director — The University of Texas at Austin
Locations (1):
- Dell Children's Medical Center, Austin, Texas, United States

IPD SHARING:
Plan to Share IPD: No
IDP will not be shared to maintain participant confidentiality.

REFERENCES:
- [Background] Spencer SP, Stoner MJ, Kelleher K, Cohen DM. Using a Multimedia Presentation to Enhance Informed Consent in a Pediatric Emergency Department. Pediatr Emerg Care. 2015 Aug;31(8):572-6. doi: 10.1097/PEC.0000000000000513. PMID 26221786
- [Background] Richardson V. Patient comprehension of informed consent. J Perioper Pract. 2013 Jan-Feb;23(1-2):26-30. doi: 10.1177/1750458913023001-204. PMID 23413533
- [Background] Sherlock A, Brownie S. Patients' recollection and understanding of informed consent: a literature review. ANZ J Surg. 2014 Apr;84(4):207-10. doi: 10.1111/ans.12555. PMID 24812707
- [Background] COMMITTEE ON BIOETHICS. Informed Consent in Decision-Making in Pediatric Practice. Pediatrics. 2016 Aug;138(2):e20161484. doi: 10.1542/peds.2016-1484. PMID 27456514
- [Background] Leazer RC. Evaluation and Management of Young Febrile Infants: An Overview of the New AAP Guideline. Pediatr Rev. 2023 Mar 1;44(3):127-138. doi: 10.1542/pir.2022-005624. PMID 36854834

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2023-09-26): https://cdn.clinicaltrials.gov/large-docs/25/NCT07074925/Prot_SAP_000.pdf